CLINICAL TRIAL: NCT06103994
Title: A Randomized, Triple-blinded, Placebo-controlled, Parallel Group Study, to Assess the Effect of Multistrain Probiotic on the Immune Response to the Influenza Vaccination
Brief Title: Study to Assess the Effect of Multistrain Probiotic on the Immune Response to the Influenza Vaccination
Acronym: LUPIN
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The Archer-Daniels-Midland Company (Industry)
Collaborators: NEXT CRO (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: CTB2022TN107
Record Dates: First submitted 2023-10-23; First posted 2023-10-27 (Actual); Last update posted 2025-04-10 (Actual); Status verified 2024-04

CONDITIONS: Influenza
Keywords: microbiome; probiotic; immune system; vaccine; influenza; flu
MeSH Terms: conditions — Influenza, Human

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Intervention (Experimental): Multistrain probiotic
  Interventions: Dietary Supplement: Multistrain probiotic
- Placebo (Placebo Comparator): Placebo
  Interventions: Other: Placebo

INTERVENTIONS:
Dietary Supplement: Multistrain probiotic — Multistrain Probiotic
  Arms: Intervention
Other: Placebo — Placebo
  Arms: Placebo

SUMMARY:
A randomized, triple-blinded, placebo-controlled, parallel group study, to assess the effect of multistrain probiotic on the immune response to the Influenza vaccination

ELIGIBILITY:
Inclusion Criteria:

1. Male or female adults aged 18-65 years
2. According to the clinical judgment of the physician, appropriate to be vaccinated against the influenza virus.
3. Able to attend study visits, comply with study requirements, and provide reliable and complete reports of AE/SAE.
4. Have been informed and have given written consent for the use of their data in accordance with local regulations before study inclusion.
5. If sexually active, commitment to use contraception methods.
6. Negative pregnancy testing (beta human chorionic gonadotropin test in urine) at V1

Exclusion Criteria:

1. Any ongoing, symptomatic acute or chronic illness requiring medical or surgical care.
2. Asymptomatic chronic conditions or findings (e.g., mild hypertension, dyslipidemia) that are not associated with evidence of end-organ damage are not exclusionary provided that they are being appropriately managed and are clinically stable (i.e., unlikely to result in symptomatic illness within the time-course of this trial) in the opinion of the investigator.
3. Acute or chronic illnesses or conditions which may be reasonably predicted to become symptomatic if treatment were withdrawn or interrupted are exclusionary, even if stable.
4. Acute or chronic illnesses reasonably expected to be associated with increased risks in the event of influenza infection (e.g., cardio-pulmonary diseases, diabetes mellitus, renal or hepatic dysfunction, hemoglobinopathies) are exclusionary, even if stable.
5. Participation in research involving a drug, biologic or device within 45 days before planned date of V2.
6. History of a serious reaction to a prior influenza vaccination (any influenza vaccine, not exclusive to INFLUVAC TETRA).
7. Hypersensitivity or allergy to INFLUVAC TETRA, its active substance, or components e.g. eggs (ovalbumin, chicken proteins), formaldehyde, cetyltrimethylammonium bromide, polysorbate 80, gentamicin, potassium chloride, potassium dihydrogen phosphate, disodium phosphate dihydrate, sodium chloride, calcium chloride dihydrate, magnesium chloride hexahydrate, water for injections.
8. Hypersensitivity or allergy to any of the ingredients of the investigational product (IP) or placebo.
9. Individuals with thrombocytopenia, any coagulation disorder or who are pharmacologically anticoagulated.
10. History of Guillain-Barré Syndrome (GBS) within 6 weeks following a previous influenza vaccine.
11. Receipt of ANY non-influenza vaccine (e.g., hepatitis B vaccine, tetanus vaccine) in the 4 weeks preceding the trial vaccination, and ANY influenza vaccine within 6 months preceding the trial vaccination, or already received the 2023-2024 influenza vaccine (any brand).
12. Planned receipt of any vaccine (other than the INFLUVAC TETRA at V2) during the study
13. Any known or suspected immunosuppressive illness, congenital or acquired, based on medical history and/or physical examination.
14. Chronic administration (defined as more than 14 continuous days) of immunosuppressants or other immune-modifying drugs within 6 months prior to the administration of the trial vaccine. An immunosuppressant dose of glucocorticoid will be defined as a systemic dose ≥ 10 mg of prednisone per day or equivalent. The use of topical, inhaled, and nasal glucocorticoids will be permitted.
15. Administration of immunoglobulins and/or any blood products within the 3 months preceding the administration of the trial vaccine or during the trial.
16. Acute disease at the time of enrolment (defined as the presence of a moderate or severe illness with or without fever, or an oral temperature >38.0°C).
17. Any condition that in the opinion of the investigator would pose a health risk to the subject if enrolled or could interfere with evaluation of the vaccine or interpretation of trial results (including neurologic or psychiatric conditions deemed likely to impair the quality of safety reporting).
18. Suspicion or recent history (within one year of planned vaccination) of alcohol or other substance abuse.
19. Smoking individuals.
20. Pregnant female, or individual who is planning on becoming pregnant during the course of the study.
21. Breastfeeding females.
22. Consumption of probiotic food supplements or use of antibiotics 1 month prior to study start.
23. Planned significant change in dietary or exercise practices during the course of the study.
24. Planned travel for more than 14 days during the course of the study.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2023-10-27 (Actual); Primary Completion 2024-01-12 (Actual); Study Completion 2024-01-12 (Actual)

PRIMARY OUTCOMES:
Change in serum strain-specific geometric mean antibody titers (determined by hemagglutination inhibition [HAI] tests) | V2 (3 weeks), V3 (6 weeks)
  Change in serum strain-specific geometric mean antibody titers (determined by hemagglutination inhibition [HAI] tests) specific for each of the 3 (out of the 4) virus strains included in the INFLUVAC TETRA vaccine, between intervention and placebo from V2 to V3. Higher values mean better immune response.

SECONDARY OUTCOMES:
Change in seroprotection rate (as measured by HAI tests) | V2 (3 weeks), V3 (6 weeks)
  Change in seroprotection rate (as measured by HAI tests) between verum and placebo groups for each of 3 (out of the 4) virus strains included in the INFLUVAC TETRA vaccine from V2 to V3. Seroprotection is defined as the proportion (percentage) of volunteers achieving an influenza antibody titer ≥1:40 by the HAI test. Higher values mean better immune response.
Change in seroconversion rate (as measured by HAI tests) | V2 (3 weeks), V3 (6 weeks)
  Change in seroconversion rate (as measured by HAI tests) between verum and placebo groups for each of 3 (out of the 4) virus strains included in the INFLUVAC TETRA vaccine from V2 to V3. Seroconversion is defined as the proportion of subjects with a pre-vaccination HAI titer <1:10 and a post-vaccination HAI titer ≥1:40 or subjects with a pre-vaccination HAI titer >1:10 and at least a 4-fold increase at day 42. Higher values mean better immune response.
Change in geometric mean neutralizing antibody (nAb) titers (as measured by microneutralization assays) | V2 (3 weeks), V3 (6 weeks)
  Change in geometric mean neutralizing antibody (nAb) titers specific for each of 3 (out of the 4) virus strains included in the INFLUVAC TETRA vaccine , as measured by a microneutralization assay from V2 to V3. Higher values mean better immune response.
Change in seroprotection rate (as measured by nAb titers in a microneutralization assay) | V2 (3 weeks), V3 (6 weeks)
  Change in seroprotection rate (as measured by nAb titers) specific for each of 3 (out of the 4) virus strains included in the INFLUVAC TETRA vaccine, as measured by a microneutralization assay from V2 to V3. Seroprotection is defined as the proportion (percentage) of volunteers achieving an influenza nAb titer ≥1:40 in MN test. Higher values mean better immune response.
Change in seroconversion rate (as measured by nAb titers in a microneutralization assay) | V2 (3 weeks), V3 (6 weeks)
  Change in seroconversion rate (as measured by nAb titers) specific for each of 3 (out of the 4) virus strains included in the INFLUVAC TETRA vaccine, as measured by a microneutralization assay from V2 to V3. Seroconversion is defined as the proportion of subjects with a pre-vaccination nAb titer <1:10 and a post-vaccination nAb titer ≥1:40 or subjects with a pre-vaccination MN titer >1:10 and at least a 4-fold increase at day 42. Higher values mean better immune response.
Change in the adaptive immune response | V2 (3 weeks), V3 (6 weeks)
  Change in the adaptive immune response, assessed by change in total plasma, strain A and B specific IgA, IgM, IgG from V2 to V3 between intervention and placebo. Higher values mean better immune response.
Change in innate immune response | V2 (3 weeks), V3 (6 weeks)
  Change in innate immune responses assessed by difference in plasma concentrations of interferon-gamma, TNF-alpha, IL-2, IL-10 from V2 to V3 between intervention and placebo. Higher values mean better immune response.
VAPI (Vaccinees' Perception of Injection) Questionnaire | V3 (6 weeks)
  VAPI (Vaccinees' Perception of Injection) Questionnaire difference at V3 between intervention and placebo. Higher values mean worse perception of the vaccine.
Change in GSRS (Gastrointestinal Symptom Rating Scale) questionnaire scoring | V1 (Baseline), V2 (3 weeks), V3 (6 weeks)
  Change in GSRS (Gastrointestinal Symptom Rating Scale) questionnaire scoring from baseline to V2,V2 to V3 and baseline to V3 between intervention and placebo. Higher values mean more troublesome symptoms
Change in stool microbiome composition | V1 (Baseline), V3 (6 weeks)
  Change in stool microbiome composition between verum and placebo between V1 and V3 in 40% of the cohort (40% of each study arm).
Adverse Events | V3 (6 weeks)
  The number of adverse events (AE)/serious adverse events (SAE) (related to the study IP) occurring during the study compared to placebo.

CONTACTS AND LOCATIONS:
Locations (1):
- Leof. Mesogeion 264,, Athens, Cholargos, Greece

IPD SHARING:
Plan to Share IPD: No